CLINICAL TRIAL: NCT02302092
Title: A Phase 3, Randomized, Double-blind, Multicenter Study Comparing the Efficacy and Safety of Intravenous Infusions of Flomoxef Versus Intravenous Infusions of Cefepime in the Treatment of Subjects With Complicated Urinary Tract Infections Including Pyelonephritis
Brief Title: An Efficacy and Safety of Flomoxef Versus Cefepime in the Treatment of Participants With Urinary Tract Infections
Acronym: FLORUS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was prematurely terminated due to administrative and strategic reasons
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLOMOXEF_301; U1111-1154-2448 (Registry Identifier: WHO)
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-06

CONDITIONS: Urinary Tract Infection
Keywords: Drug Therapy
MeSH Terms: conditions — Urinary Tract Infections | interventions — flomoxef; Cefepime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flomoxef (Experimental): Flomoxef, 2g, injection, intravenously, twice daily (every 12 hours), for up to 12 days.
  Interventions: Drug: Flomoxef
- Cefepime (Active Comparator): Cefepime, 1g, injection, intravenously, twice daily (every 12 hours) for up to 14 days.
  Interventions: Drug: Cefepime

INTERVENTIONS:
Drug: Flomoxef — Flomoxef intravenous infusion
  Arms: Flomoxef
Drug: Cefepime — Cefepime intravenous infusion
  Other Names: Maxipime
  Arms: Cefepime

SUMMARY:
The purpose of this study is to compare the effectiveness of antibiotic flomoxef with cefepime for the treatment of complicated urinary tract infections (cUTIs) in Russian adults.

DETAILED DESCRIPTION:
The drug being tested in this study is called Flomoxef. Flomoxef is being tested in people with a complicated urinary tract infection (cUTI) including a kidney infection. This study compares Flomoxef to Cefepime, another antibiotic.

The study enrolled 13 patients.

Participants are randomly assigned by a computer generated number to one of two treatment groups:

* Flomoxef - intravenous infusion 2g twice daily (every 12 hours); or
* Cefepime - intravenous infusion 1g twice daily (every 12 hours).

This multi-center trial is conducted at 4 sites in the Russian Federation. The overall time to participate in this study is 30+/-3 days. Participants make six visits to the clinic.

Study was prematurely terminated due to administrative and strategic reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Is a man or woman aged 18 to 70 years, inclusive.
2. Has pyuria (a white blood cell [WBC] count greater than 10/μL in unspun urine or greater than or equal to 10 per high power field in spun urine).
3. Has clinical signs and/or symptoms of a complicated lower urinary tract infection (UTI) and/or acute pyelonephritis that include one or more of the following: fever (i.e, axillary temperature greater than 37.7°C), chills, malaise, flank pain, back pain, and/or costo-vertebral angle pain or tenderness and/or any symptoms of dysuria (dysuria, urinary urgency, urinary frequency, suprapubic discomfort, new urinary incontinence or worsening of pre-existing incontinence) that occur in the presence of a functional or anatomical abnormality of the urinary tract or in the presence of catheterization.
4. Has a pretreatment baseline urine culture specimen obtained within 24 hours before the administration of the first dose of study drug (NOTE: Participants may be enrolled in this study and start intravenous (IV) study drug therapy before the Investigator knows the results of the baseline urine culture).
5. Requires IV antibacterial therapy for the treatment of the presumed complicated UTI (cUTI).
6. In the opinion of the investigator, is capable of understanding and complying with protocol requirements.
7. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures, or has a legally acceptable representative sign the forms.
8. Meets protocol-specified criteria regarding the use of contraception; and 9-Is willing and able to comply with study procedures.

Exclusion Criteria:

1. Has received any investigational compound within 30 days of screening.
2. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, or sibling) or may consent under duress.
3. Is a female participant who is pregnant or lactating or intending to become pregnant before, during, or within one month after participating in this study, or intends to donate ova during such time period.
4. Is a male participant who intends to donate sperm during the course of this study or for 12 weeks thereafter.
5. Has participated in another clinical study within the past 30 days.
6. Has a history of allergy to or intolerance of beta-lactams (penicillins, cephalosporins or carbopenems).
7. Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise: 1) the safety or well-being of the participant or study staff, 2) the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding), or 3) the analysis of results.
8. Has received any amount of potentially therapeutic antibacterial therapy after collection of the pretreatment baseline urine culture and before administration of the first dose of study drug.
9. Has received any dose of a potentially therapeutic antibacterial agent for the treatment of the current UTI within 48 hours before providing the pretreatment baseline urine culture specimen.
10. Has a current urinary catheter that is not scheduled to be removed before the End-of-Therapy (EOT) visit (intermittent straight catheterization during the IV study drug administration period is acceptable).
11. Has any history of trauma to the pelvis or urinary tract within one year before the screening visit.
12. Has any other contraindications to the medicines that are to be used in the study (according to the manufacturer's instructions).
13. Is considered unlikely to survive the four-week study period or has any rapidly progressing disease or immediately life-threatening illness (including acute hepatic failure, respiratory failure or septic shock).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-02-02 (Actual); Study Completion 2016-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (5):
- Russia (5):
  - Moscow
  - Rostov-on-Don
  - Saint Petersburg
  - Volgograd
  - Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in Russia from 01 December 2015 to 15 Feb 2016.
Pre-assignment Details: Participants with a diagnosis of complicated urinary tract infections were enrolled in 1:1 ratio to flomoxef or cefepime arm groups.
Groups:
- Flomoxef: Flomoxef, 2g, injection, intravenously, twice daily (every 12 hours) for up to 12 days.
Period: Overall Study
Arm/Group | Flomoxef | Cefepime
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population included all participants who received any dose of planned study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Flomoxef | Cefepime | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (17.1) | 53.3 (12.9) | 54.1 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Russia | 6 | 7 | 13
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2].
  kg/m^2 | 25.443 (4.821) | 31.041 (8.321) | 28.458 (7.262)
Smoking status [Number; unit: participants]
  Non-tobacco user | 4 | 6 | 10
  Tobacco user | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Resolution of All Clinical Symptoms of a Complicated Urinary Tract Infection (cUTI) at the End of Treatment (EOT) Visit
Description: At the EOT visit (Days 7 to 14), the Investigator collected information about each symptom and performed a judgement about the participant's status. Clinical symptoms present at trial entry were considered to be resolved if the participant has no pyuria; no fever; no malaise, flank pain, back pain, and/or costo-vertebral angle pain or tenderness; and no symptoms of dysuria, urinary urgency, urinary frequency, suprapubic discomfort, new urinary incontinence, or worsening of pre-existing incontinence. Resolution of all clinical symptoms of cUTI were assessed relative to baseline.
Time Frame: Baseline and Days 7 to 14
Population: The micro-intent to treat (ITT) population included all participants who were randomized and had a baseline bacterial pathogen on culture of urine that causes UTI against which the investigational drug has antibacterial activity.
Measure: Number; unit: percentage of participants
Arm/Group | Flomoxef | Cefepime
Number analyzed (Participants) | 5 | 7
percentage of participants | 60.0 | 42.9

2. Secondary Outcome: Percentage of Participants With Microbiological Success at the EOT and Test-of-Cure (TOC) Visits
Description: A urine sample was collected at EOT (Days 7 to 14) and TOC (Days 14 to 21) visits to determine level of uropathogen. Cultures of urine sample were processed by calibrated loop to identify a quantitative count of bacteria, with a lower limit of 10^4 colony forming units per milliliter (CFU/mL). Microbiological success was defined as bacterial uropathogen level of <10^4 CFU/mL. Microbiological response was categorized as:microbiological eradication/persistence/new infection/superinfection. An infection was eradicated if all uropathogens isolated at study entry at a level ≥10^4 CFU/mL have decreased to <10^4 CFU/mL, persistent if level of uropathogen has increased by ≥10^4 CFU/Ml. A new infection, if there is isolation and growth of a uropathogen other than original pathogen and superinfection if there is growth of a uropathogen other than original pathogen at a level ≥10^4 CFU/mL. Microbiological success was assessed relative to baseline.
Time Frame: Baseline, Days 7 to 14 and 14 to 21
Population: The micro-ITT population included all participants who were randomized and had a baseline bacterial pathogen on culture of urine that causes UTI against which the investigational drug has antibacterial activity.
Measure: Number; unit: percentage of participants
Arm/Group | Flomoxef | Cefepime
Number analyzed (Participants) | 5 | 7
percentage of participants
  Days 7 to 14: Eradication | 80.0 | 85.7
  Days 7 to 14: New infection | 0.0 | 14.3
  Days 7 to 14: Persistence | 20.0 | 14.3
  Days 7 to 14: Superinfection | 0.0 | 14.3
  Days 14 to 21: Eradication | 80.0 | 85.7
  Days 14 to 21: New infection | 20.0 | 14.3
  Days 14 to 21: Persistence | 0.0 | 14.3
  Days 14 to 21: Superinfection | 40.0 | 28.6

3. Secondary Outcome: Percentage of Participants Who Achieved Clinical Resolution of Symptoms of a cUTI at Visit 3, TOC and Late Follow-up (LFU) Visits
Description: At Visit 3 (Day 3) and at the TOC (Days 14 to 21) and LFU visits (Day 30), the Investigator collected information about each symptom and performed a judgement about the participant's status. Clinical symptoms present at trial entry were considered to be resolved if the participant has no pyuria; no fever; no malaise, flank pain, back pain, and/or costo-vertebral angle pain or tenderness; and no symptoms of dysuria, urinary urgency, urinary frequency, suprapubic discomfort, new urinary incontinence, or worsening of pre-existing incontinence. Resolution of all clinical symptoms of cUTI were assessed relative to baseline.
Time Frame: Baseline, Days 3, 14 to 21 and 30
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Flomoxef | Cefepime
Number analyzed (Participants) | 5 | 7
percentage of participants
  Day 3 | 0.0 | 14.3
  Days 14 to 21 | 60.0 | 28.6
  Day 30 | 60.0 | 57.1

4. Secondary Outcome: Percentage of Participants With Microbiologic Eradication of the Unique Pathogen at the EOT and TOC Visits
Description: A urine sample was collected from the participants at the EOT (Days 7 to 14) and TOC (Day 14 to 21) visits to determine the level of uropathogen. Cultures of the urine sample were processed by using a calibrated loop to identify a quantitative count of bacteria, with a lower limit of 10^4 CFU/mL. Microbiological response at the TOC visit was based on the same grades as for the EOT visit. The infection was considered to be eradicated if all uropathogens isolated at study entry at a level equal to or greater than 10^4 CFU/mL have decreased to less than 10^4 CFU/mL.
Time Frame: Baseline, Days 7 to 14 and 14 to 21
Population: Due to premature trial termination and small sample size, data for eradication for particular pathogen numbers in different time periods was not determined.
Arm/Group | Flomoxef | Cefepime
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Microbiologic Persistence of the Unique Pathogen at the EOT and TOC Visits
Description: A urine sample was collected from the participants at the EOT (Days 7 to 14) and TOC (Days 14 to 21) visits to determine the level of uropathogen. Cultures of the urine sample was processed by using a calibrated loop to identify a quantitative count of bacteria, with a lower limit of 10^4 CFU/mL. Microbiological response at the TOC visit was be based on the same grades as for the EOT visit. The infection was considered to be persistent if the level of the uropathogen has increased by greater than or equal to 10^4 CFU/mL from the time of study entry to that of the EOT and TOC visits.
Time Frame: Baseline, Days 7 to 14 and 14 to 21
Population: Due to premature trial termination and small sample size, data for persistence of particular pathogen numbers in different time periods was not determined.
Arm/Group | Flomoxef | Cefepime
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With a New Infection at the EOT and TOC Visits
Description: A urine sample was collected from the participants at the EOT (Days 7 to 14) and TOC (Days 14 to 21) visits to determine the level of uropathogen. Cultures of the urine sample were processed by using a calibrated loop to identify a quantitative count of bacteria, with a lower limit of 10^4 CFU/mL. A new infection was defined as the isolation and growth of a uropathogen other than the original pathogen.
Time Frame: Baseline, Days 7 to 14 and 14 to 21
Population: Due to premature trial termination and small sample size, data for new infection due to particular pathogen numbers in different time periods was not determined.
Arm/Group | Flomoxef | Cefepime
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With a Superinfection at the EOT and TOC Visits
Description: A urine sample was collected from the participants at the EOT (Days 7 to 14) and TOC (Days 14 to 21) visits to determine the level of uropathogen. Cultures of the urine sample were processed by using a calibrated loop to identify a quantitative count of bacteria, with a lower limit of 10^4 CFU/mL. A superinfection was defined as growth of a uropathogen other than the original pathogen at a level greater than or equal to 10^4 CFU/mL at any time during the course of active therapy.
Time Frame: Baseline, Day 7 to 14 and 14 to 21
Population: Due to premature trial termination and small sample size, data for superinfection due to particular pathogen numbers in different time periods was not determined.
Arm/Group | Flomoxef | Cefepime
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Treatment-Emergent-Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A Serious Adverse Event (SAE) A serious is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: Baseline up to Day 30
Population: The safety population included all participants who received any dose of planned study medication.
Measure: Number; unit: participants
Arm/Group | Flomoxef | Cefepime
Number analyzed (Participants) | 6 | 7
participants
  SAEs | 0 | 0
  TEAEs | 2 | 2

9. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Values
Description: The number of participants with any markedly abnormal (above or below normal ranges) standard safety laboratory values was collected throughout study.
Time Frame: Day 21
Population: The safety population included all participants who received any dose of planned study medication.
Measure: Number; unit: participants
Arm/Group | Flomoxef | Cefepime
Number analyzed (Participants) | 6 | 7
participants
  Neutrophil count decreased | 1 | 0
  White blood cells count increased | 1 | 0
  C-reactive Protein level increased | 1 | 0
  C-reactive Protein level decreased | 0 | 1

10. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Signs
Description: Vital signs included body temperature (axillary measurement), diastolic and systolic blood pressure (5 minutes), respiratory rate, and pulse (bpm).
Time Frame: Day 1 up to Day 21
Population: The safety population included all participants who received any dose of planned study medication.
Measure: Number; unit: participants
Arm/Group | Flomoxef | Cefepime
Number analyzed (Participants) | 6 | 7
participants
  Day 1: Systolic Blood Pressure | 0 | 0
  Day 3: Systolic Blood Pressure | 0 | 0
  Day 7-14: Systolic Blood Pressure | 0 | 0
  Day 14-21: Systolic Blood Pressure | 0 | 0
  Day 1: Diastolic Blood Pressure | 0 | 0
  Day 3: Diastolic Blood Pressure | 0 | 0
  Day 7-14: Diastolic Blood Pressure | 0 | 0
  Day 14-21: Diastolic Blood Pressure | 0 | 0
  Day 1: Pulse Rate | 0 | 0
  Day 3: Pulse Rate | 0 | 0
  Day 7-14: Pulse Rate | 0 | 0
  Day 14-21: Pulse Rate | 0 | 0
  Day 1: Respiration Rate | 0 | 0
  Day 3: Respiration Rate | 0 | 0
  Day 7-14: Respiration Rate | 0 | 0
  Day 14-21: Respiration Rate | 0 | 0
  Day 1: Body Temperature | 2 | 2
  Day 3: Body Temperature | 0 | 0
  Day 7-14: Body Temperature | 0 | 0
  Day 14-21: Body Temperature | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Change in Physical Examination Findings
Description: Physical examination consists of examinations of the following body systems: (1) cardiovascular system; (2) dermatologic system (3) ears, nose, throat; (4) extremities; (5) eyes; (6) gastrointestinal system; (7) genitourinary system; (8) lymph nodes; (9) musculoskeletal system; (10) nervous system; (11) respiratory system.
Time Frame: Day 1 up to Day 21
Population: The safety population included all participants who received any dose of planned study medication.
Measure: Number; unit: participants
Arm/Group | Flomoxef | Cefepime
Number analyzed (Participants) | 6 | 7
participants
  Day 1: Cardiovascular system | 0 | 0
  Day 3: Cardiovascular system | 0 | 0
  Day 7-14: Cardiovascular system | 1 | 0
  Day 14-21: Cardiovascular system | 1 | 0
  Day 1: Dermatologic system | 0 | 0
  Day 3: Dermatologic system | 0 | 0
  Day 7-14: Dermatologic system | 0 | 0
  Day 14-21: Dermatologic system | 0 | 0
  Day 1: Ear/Nose/Tongue | 0 | 0
  Day 3: Ear/Nose/Tongue | 0 | 0
  Day 7-14: Ear/Nose/Tongue | 0 | 0
  Day 14-21: Ear/Nose/Tongue | 0 | 0
  Day 1: Extremities | 0 | 0
  Day 3: Extremities | 0 | 0
  Day 7-14: Extremities | 0 | 0
  Day 14-21: Extremities | 0 | 0
  Day 1: Eyes | 0 | 0
  Day 3: Eyes | 0 | 0
  Day 7-14: Eyes | 0 | 0
  Day 4-21: Eyes | 0 | 0
  Day 1: Gastrointestinal system | 0 | 0
  Day 3: Gastrointestinal system | 0 | 0
  Day 7-14: Gastrointestinal system | 0 | 0
  Day 14-21: Gastrointestinal system | 0 | 0
  Day 1: Genitourinary system | 6 | 7
  Day 3: Genitourinary system | 3 | 6
  Day 7-14: Genitourinary system | 0 | 1
  Day 14-21: Genitourinary system | 0 | 1
  Day 1: Lymph nodes | 0 | 0
  Day 3: Lymph nodes | 0 | 0
  Day 7-14: Lymph nodes | 0 | 0
  Day 14-21: Lymph nodes | 0 | 0
  Day 1: Musculoskeletal system | 0 | 0
  Day 3: Musculoskeletal system | 0 | 0
  Day 7-14: Musculoskeletal system | 0 | 0
  Day 14-21: Musculoskeletal system | 0 | 0
  Day 1: Nervous system | 0 | 0
  Day 3: Nervous system | 0 | 0
  Day 7-14: Nervous system | 0 | 0
  Day 14-21: Nervous system | 0 | 0
  Day 1: Respiratory system | 0 | 0
  Day 3: Respiratory system | 0 | 0
  Day 7-14: Respiratory system | 0 | 0
  Day 14-21: Respiratory system | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 30
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Flomoxef | Cefepime
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 2/6 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flomoxef (N=6) | Cefepime (N=7)
Pyrexia (General disorders) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study is limited as only 13 out of the original 80 participants planned entered the study, due to this none of the planned statistical analyses from the protocol could be carried out, and all results should be reviewed with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.